CLINICAL TRIAL: NCT07296393
Title: The Association Between Umbilical Cord Blood Vitamin A Levels and Adverse Outcomes in Extremely Preterm Infants: A Single-Center Prospective Cohort Study
Brief Title: Vitamin A in Cord Blood and Preterm Outcomes
Status: Not yet recruiting | Type: Observational
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Sponsor
Other Study IDs: 25K281-001
Record Dates: First submitted 2025-12-09; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Extremely Premature Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Extremely Preterm Infants

SUMMARY:
This single-center prospective cohort study aims to describe the distribution of umbilical-cord blood vitamin A concentrations in extremely preterm infants (<32 weeks' gestation) and to evaluate whether low cord blood vitamin A is associated with increased risk of neonatal morbidities such as bronchopulmonary dysplasia (BPD), necrotising enterocolitis (NEC), severe intraventricular haemorrhage (IVH), retinopathy of prematurity (ROP), periventricular leukomalacia (PVL), high-grade patent ductus arteriosus (hsPDA), respiratory distress syndrome (RDS), sepsis and death before discharge.

ELIGIBILITY:
Inclusion Criteria:

Gestational age <32 weeks Birth at First Hospital of Jilin University Umbilical cord blood sample obtained within 24 h Parental written informed consent

Exclusion Criteria:

Major congenital malformation or chromosomal abnormality Refusal of consent

Max Age: 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preterm neonates (gestational age <32 weeks)
Sampling Method: Probability Sample
Enrollment: 155 (Estimated)
Dates: Start 2025-12-10 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Composite adverse neonatal outcome (any of death, moderate-severe BPD, NEC≥stage II, IVH≥grade III, ROP≥stage 3, PVL, hsPDA, culture-proven sepsis) | From birth to 36 weeks' PMA or discharge, up to 3 months chronological age.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Allen LH, Miller JW, de Groot L, Rosenberg IH, Smith AD, Refsum H, Raiten DJ. Biomarkers of Nutrition for Development (BOND): Vitamin B-12 Review. J Nutr. 2018 Dec 1;148(suppl_4):1995S-2027S. doi: 10.1093/jn/nxy201. PMID 30500928